CLINICAL TRIAL: NCT01228175
Title: Effectiveness of Varenicline: Testing Individual Differences
Acronym: Varenicline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kent Hutchison, Ph.D., Chief Science Officer, The Mind Research Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01DA025074 (NIH); R01DA025074 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-10-26 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Smoking Addiction
MeSH Terms: interventions — Riboflavin; Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): Varenicline
  Interventions: Drug: Varenicline
- Microcrystal Cellulose (Placebo Comparator): Microcrystal cellulose placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 25mg look alike riboflavin tablets to match active study medication.
  Other Names: riboflavin
  Arms: Microcrystal Cellulose
Drug: Varenicline — Days 1-3 - .5mg tablet 1xdaily Days 4-7 - .5mg tablet 2xdaily Days 8-84 - 1mg tablet 2xdaily
  Other Names: Chantix
  Arms: Varenicline

SUMMARY:
The study will evaluate the effectiveness of smoking cessation using Varenicline versus placebo. Effectiveness will be measured by the average number of cigarettes smoked per smoking day for up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs to 55 yrs
* smoker

Exclusion Criteria:

* Medical Contraindications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2010-03; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hutchison, Ph.D, Principal Investigator — Director, Neurogenetics Core, The Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Microcrystal Cellulose
Started | 119 | 99
Completed | 53 | 46
Not Completed | 66 | 53
Not completed — Lost to Follow-up | 64 | 50
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Microcrystal Cellulose | Total
Number analyzed (Participants) | 119 | 99 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 99 | 218
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 64 | 145
  Male | 38 | 35 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 119 | 99 | 218

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Smoking Day
Description: The number of cigarettes smoked were assessed only on a "smoking day", i.e., when a participant smoked at least 1 cigarette. Data was recorded each day for up to 36 weeks.
Time Frame: up to 36 weeks
Measure: Mean (Standard Deviation); unit: Cigarettes per smoking day
Arm/Group | Varenicline | Microcrystal Cellulose
Number analyzed (Participants) | 53 | 46
Cigarettes per smoking day | 4.9256 (5.62357) | 8.4989 (8.53172)

ADVERSE EVENTS:
Arm/Group | Varenicline | Microcrystal Cellulose
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/99
Other Adverse Events (participants affected / at risk) | 0/119 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No